CLINICAL TRIAL: NCT02331862
Title: To Study the Effect of Adjunctive Oral Methylprednisolone Therapy in Pediatric Urinary Tract Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-103-050
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Urinary Tract Infection
Keywords: urinary tract infection; methylprednisolone
MeSH Terms: conditions — Urinary Tract Infections | interventions — Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UTI treated with Methylprednisolone (Experimental): UTI treated with Methylprednisolone in addition to the effective antibiotics
  Interventions: Drug: Methylprednisolone
- UTI not treated with Methylprednisolone (No Intervention): UTI treated with effective antibiotics only

INTERVENTIONS:
Drug: Methylprednisolone — Add methylprednisolone in addition to the experience antibiotics in children with urinary tract infection to see if the frequency of the renal scar formation could be decreased
  Other Names: Adrenal corticosteroid
  Arms: UTI treated with Methylprednisolone

SUMMARY:
Purposes of this study will be as follows:

1. To design a prospective, randomized, and open-labeled study to investigate the effect and the side effect of MPD in combination with conventional antibiotics to affect clinical course, outcome, and medical expenses.
2. To compare level of the urinary and serum cytokines before and after received MPD for the following sub-aim:

I. To determine the population who is benefit from MPD to reduce the severity of clinical course and subsequent renal scarring.

II. To understand the mechanism by which the MPD could shorten the clinical course and reduce the renal scarring.

DETAILED DESCRIPTION:
The urinary tract infection (UTI) is a common etiology of the febrile children and the acute pyelonephritis (APN) happen in 70% children with the first febrile UTI. After the first APN, the irreversible renal scarring takes place in about 40% patients. The sequela of the renal scarring includes chronic kidney disease, hypertension, the complication during the pregnancy, and even the end stage of renal diseases. Due to the progression of the pathophysiology of the pyelonephritis and the renal scarring in the past years, we understand that the inflammation is one of the important mechanisms. Therefore, there are many animal studies clarifying the role of the anti-inflammation or antioxidant to reduce the renal scarring. In our previous studies, Dr. Chiou Y.Y. and colleagues has provided the evidence that the adjunctive methylprednisolone (MPD) can decrease the risk of the renal scarring for patients with high risk APN, which was defined as inflammatory volume more than 4.6 mL on technetium-99m-labeled dimercaptosuccinic acid scan or abnormal renal ultrasonography results. Our study is the first human study demonstrating the solution for the renal scarring. However, whether this result can be applied to the whole spectrum of the UTI is still unknown. Purposes of this study will be as follows:

1. To design a prospective, randomized, and open-labeled study to investigate the effect and the side effect of MPD in combination with conventional antibiotics to affect clinical course, outcome, and medical expenses.
2. To compare level of the urinary and serum cytokines before and after received MPD for the following sub-aim:

I. To determine the population who is benefit from MPD to reduce the severity of clinical course and subsequent renal scarring.

II. To understand the mechanism by which the MPD could shorten the clinical course and reduce the renal scarring.

According to these studies, we will provide a new and effective guideline to shorten disease course, save medical expenses, and decrease the risk for renal scarring sequela.

ELIGIBILITY:
Inclusion Criteria:

* 1week old ~ 16 years old children with UTI

Exclusion Criteria:

* Previous UTI
* Known GU tract obstruction
* Severe sepsis with vital signs change
* Antibiotics used

Ages: 1 Week to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with renal scar formation | 6.5 months
  Check the renal scar formation 6.5 months after the UTI

SECONDARY OUTCOMES:
Duration of the hospitalization | the duration patient in the hospital, may be about 5 days
  Check the duration of the hospitalization
Expense of the hospitalization | the duration patient in the hospital, may be about 5 days
  Check the expense of the hospitalization